CLINICAL TRIAL: NCT01982487
Title: A Phase I/IIb Study of Recombinant ALVAC(2)-NY-ESO-1 (M)/TRICOM in Combination With INCB024360 for Patients in Remission With Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma Whose Tumors Express NY-ESO-1 or LAGE-1 Antigen
Brief Title: Vaccine Therapy and IDO1 Inhibitor INCB024360 in Treating Patients With Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Are in Remission
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 243013; NCI-2013-02080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 080913; SRC1 082013; IRB 100313; SRC2 082713; I 243013 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer; Stage IA Fallopian Tube Cancer; Stage IA Ovarian Epithelial Cancer; Stage IA Primary Peritoneal Cavity Cancer; Stage IB Fallopian Tube Cancer; Stage IB Ovarian Epithelial Cancer; Stage IB Primary Peritoneal Cavity Cancer; Stage IC Fallopian Tube Cancer; Stage IC Ovarian Epithelial Cancer; Stage IC Primary Peritoneal Cavity Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Epithelial Cancer; Stage IIA Primary Peritoneal Cavity Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Epithelial Cancer; Stage IIB Primary Peritoneal Cavity Cancer; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Epithelial Cancer; Stage IIC Primary Peritoneal Cavity Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Primary Peritoneal Cavity Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Primary Peritoneal Cavity Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Primary Peritoneal Cavity Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (no treatment) (No Intervention): Patients receive no treatment.
- Arm B (IDO1 inhibitor INCB024360) (Experimental): Patients receive IDO1 inhibitor INCB024360 PO BID on days 1-28.
  Interventions: Drug: IDO1 inhibitor INCB024360; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm C (vaccine, IDO1 inhibitor INCB024360) (Experimental): Patients receive ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine SC on day 1 and IDO1 inhibitor INCB024360 PO BID on days 1-28.
  Interventions: Biological: ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine; Drug: IDO1 inhibitor INCB024360; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm D (vaccine) (Experimental): Patients receive ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine SC on day 1.
  Interventions: Biological: ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine — Given SC
  Other Names: vCP2292
  Arms: Arm C (vaccine, IDO1 inhibitor INCB024360); Arm D (vaccine)
Drug: IDO1 inhibitor INCB024360 — Given PO
  Other Names: INCB024360; indoleamine-2,3-dioxygenase inhibitor INCB024360
  Arms: Arm B (IDO1 inhibitor INCB024360); Arm C (vaccine, IDO1 inhibitor INCB024360)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm B (IDO1 inhibitor INCB024360); Arm C (vaccine, IDO1 inhibitor INCB024360); Arm D (vaccine)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
  Arms: Arm B (IDO1 inhibitor INCB024360); Arm C (vaccine, IDO1 inhibitor INCB024360); Arm D (vaccine)

SUMMARY:
This partially randomized phase I/IIb trial studies the side effects vaccine therapy and indoleamine 2,3-dioxygenase (IDO1) inhibitor 4-amino-1,2,5-oxadizaole-3-carboximidamide (INCB024360) and to see how well they work in treating patients with epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in remission. Vaccines made from gene-modified virus may help the body build an effective immune response to kill tumor cells. IDO1 inhibitor INCB024360 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vaccine therapy with IDO1 inhibitor INCB024360 may be an effective treatment for epithelial ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of fixed doses of the modified canarypox vector (ALVAC[2])-cancer/testis antigen 1B (NY-ESO-1) (M)/triad of costimulatory molecules (TRICOM) vaccine in combination with INCB024360 (IDO1 inhibitor INCB024360). (Phase I) II. To evaluate toxicity as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. (Phase I) III. To determine the progression free survival (PFS) using standard imaging response (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) criteria. (Phase IIb)

SECONDARY OBJECTIVES:

I. To determine the effectiveness of INCB024360 on enhancing vaccine efficacy by assessing NY-ESO-1 specific cellular and humoral immunity in peripheral blood NY-ESO-1 specific CD8+ and CD4+ T cells.

II. To determine the effectiveness of INCB024360 on enhancing vaccine efficacy by assessing NY-ESO-1 specific cellular and humoral immunity in peripheral blood NY-ESO-1 specific antibodies.

III. To determine the effectiveness of INCB024360 on enhancing vaccine efficacy by assessing NY-ESO-1 specific cellular and humoral immunity in peripheral blood frequency of CD4+CD25+FOXP3+ regulatory T cells.

IV. To determine the effectiveness of INCB024360 on enhancing vaccine efficacy by assessing NY-ESO-1 specific cellular and humoral immunity in pharmacokinetics (PK) of IDO in relation to T cell frequency and function in correlation with PFS.

OUTLINE: This is a Phase I study followed by a randomized Phase IIb study.

PHASE I: Patients receive ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine subcutaneously (SC) on day 1 and IDO1 inhibitor INCB024360 orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

PHASE IIb: Patients are randomized to 1 of 4 arms.

ARM A: Patients receive no treatment.

ARM B: Patients receive IDO1 inhibitor INCB024360 PO BID on days 1-28.

ARM C: Patients receive ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine SC on day 1 and IDO1 inhibitor INCB024360 PO BID on days 1-28.

ARM D: Patients receive ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine SC on day 1.

In all arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 weeks; at 3, 6, and 12 months; and then annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with epithelial ovarian, fallopian tube, or primary peritoneal carcinoma and no evidence of disease or no measurable disease after 1st or 2nd line therapy; these patients would normally enter a period of observation after standard management
* Any human leukocyte antigen (HLA) type; historic HLA typing is permitted
* Tumor expression of NY-ESO-1 or cancer/testis antigen 2 (LAGE-1) by immunohistochemistry (IHC) and/or reverse transcription-polymerase chain reaction (RTPCR)
* No allergy to eggs
* Life expectancy > 6 months
* Hematology and biochemistry laboratory results within the limits normally expected for the patient population, without evidence of major organ failure
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelet count (PLT) >= 75,000/uL
* Hemoglobin (Hgb) >= 8g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum aspartate aminotransferase (serum glutamic oxalacetic transaminase [SGOT]/aspartate aminotransferase [AST]) or serum alanine aminotransferase (serum glutamate pyruvate transaminase [SGPT]/alanine aminotransferase [ALT]) =< 3 x ULN
* Serum creatinine =< 2 x ULN
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5
* Have been informed of other treatment options
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* The ability to swallow and retain oral medication
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patients may have received previous NY-ESO-1 vaccine therapy; patients who received maintenance paclitaxel or bevacizumab are eligible for enrollment provided they have discontinued therapy (at least 4 weeks for prior taxane) prior to randomization and recovered from toxicities to less than grade 2

Exclusion Criteria:

* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available
* Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders)
* History of autoimmune disease (e.g. thyroiditis, lupus) except vitiligo
* Concomitant systemic treatment with corticosteroids, anti-histamine or non-steroidal anti-inflammatory drugs, and other platelet inhibitory agents
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing of study drug (6 weeks for nitrosoureas); concomitant hormonal therapies for breast cancers are allowed
* Clinically significant heart disease (New York Heart Association [NYHA] class III or class IV) within 6 months
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study drug
* Known hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of availability of a patient for immunological and clinical follow-up assessment
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the investigator's opinion will prevent completion of the protocol therapy or follow-up
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug (i.e., any significant medical illness or abnormal laboratory finding that would, in the investigator's judgement, increase the patient's risk by participating in this study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of IDO1 inhibitor INCB024360, determined by incidence of dose limiting toxicities graded according to the NCI CTCAE version 4.0 (Phase I) | 28 days
PFS (Phase IIb) | Up to 15 years
  The primary analysis will be carried forth using a Cox proportional hazards model with factors corresponding to treatment combination, IDO1 inhibitor INCB024360 (yes/no) and ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine (yes/no), a continuous covariate adjustment for the length of the treatment free interval and a blocking factor.

SECONDARY OUTCOMES:
Immunological response | Up to 12 months
  Immunological parameters (antibody titres, NY-ESO-1 specific CD8+ and CD4+ frequency and function, frequency of memory T cell populations, TCR avidity, secondary recall response) will be analyzed in a straightforward analysis-of-covariance (ANCOVA) fashion modeling post-treatment levels as a function of pre-treatment levels with factors corresponding to IDO1 inhibitor INCB024360 (yes/no) and ALVAC(2)-NY-ESO-1 (M)/TRICOM vaccine (yes/no).
Toxicity rate, graded according to NCI CTCAE version 4.0 | Up to 12 months
  The toxicity rate will be estimated using a one-sided, 95%, exact binomial confidence interval (Clopper-Pearson). The lower one sided limit will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, Principal Investigator — Roswell Park Cancer Institute